CLINICAL TRIAL: NCT04095728
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Study Investigating the Efficacy of Brain Octane® Oil (Caprylic Acid Triglycerides) on Cognition, Coordination, Reaction Time and Measurements of Physical Performance in Recreationally Active Adults
Brief Title: Investigating the Efficacy of Brain Octane® Oil on Cognition, Coordination, Reaction Time and Measurements of Physical Performance in Recreationally Active Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulletproof 360, Inc. (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 19BCHB
Record Dates: First submitted 2019-09-16; First posted 2019-09-19 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: Cognition; Healthy; Brain Octane Oil; Caprylic acid triglycerides; Physical performance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Product (Experimental)
  Interventions: Dietary Supplement: Brain Octane Oil
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Brain Octane Oil — Participants will complete a 7-day dose escalation period, and then consume 2 servings of the study product (1 serving = 1 tablespoon) for 21 days.
  Other Names: caprylic acid triglycerides
  Arms: Investigational Product
Other: Placebo — Participants will complete a 7-day dose escalation period, and then consume 2 servings of the study product (1 serving = 1 tablespoon) for 21 days.
  Other Names: High Oleic Sunflower Oil
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel study investigating the efficacy of Brain Octane® Oil on cognition, coordination, reaction time and measurements of physical performance in recreationally active adults. Thirty eligible participants will consume the investigational product or placebo for 27 days. 15 participants will consume the investigational product and 15 participants will receive the placebo product to consume.

The primary outcome is assessing reaction time, cognition, and the ability to perform cognitive tasks. Assessments will be conducted at baseline, and end of study (30 days apart).

ELIGIBILITY:
Inclusion Criteria:

1. Provided voluntary, written, informed consent to participate in the study.
2. Males and females between ages 25-55 years old inclusive
3. Body mass index (BMI) in the range of 19.0 and 29.9 kg/m2 inclusive
4. Female participants not of child-bearing potential, defined as females who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, total endometrial ablation) or have been post-menopausal (natural or surgically) for at least 1 year prior to screening

   Or,

   Females of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
5. Athletes engaging in endurance exercise (examples include but are not limited to running, cycling, swimming, and skiing) at least 1x per week for a weekly total of at least 1-hour
6. Good general health to perform exercise testing safely, as determined by the Qualified Investigator based on medical history, physical examination, ECG and laboratory results
7. Healthy as determined by laboratory results, medical history, and physical exam by the Qualified Investigator (QI)
8. Willingness to complete questionnaires, records, and diaries associated with the study and to complete all study procedures at all clinic visits
9. Agrees to maintain their normal dietary pattern and exercise routine throughout the study
10. Agrees to maintain their daily caloric intake by adjusting their normal diet to account for the additional 250 calories from the Brain Octane® Oil

Exclusion Criteria:

1. Women who are pregnant, breast feeding, or planning to become pregnant during the course of the trial
2. Known allergy to the test material's active or inactive ingredients
3. Abnormal respiratory function (examples include but are not limited to asthma, exercise-induced asthma, exercise-induced respiratory problems) that in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant.
4. Visual impairment that limits the ability to perform study assessments
5. Cancer, except skin cancers completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
6. Blood/bleeding disorders with the exception of a history of anemia caused by a deficiency of a mineral or vitamin, and no longer present
7. Clinically significant abnormal laboratory results at screening as determined by the QI.
8. Any autoimmune disease or immune-compromised (i.e. HIV positive, use of anti-rejection medication, rheumatoid arthritis, etc.)
9. Verbal confirmation of the diagnosis of Hepatitis B/C positive
10. Verbal confirmation of current or pre-existing thyroid condition except for hypothyroidism that has been treated with a stable dose of medication for at least 6 months
11. Cardiac diseases that in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant.
12. Liver or renal conditions (e.g. cirrhosis of the liver, kidney disease, etc.) that in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant. Asymptomatic kidney stones are allowed.
13. Current oral or gastrointestinal pathology (e.g. mouth ulcers, chronic diarrhea, inflammatory bowel disease, uncontrolled GERD), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), or other conditions known to interfere with the absorption, distribution, metabolism or excretion
14. History of or current diagnosis of Type I or Type II diabetes
15. Presence or history of neurological disorders or significant psychiatric illness that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant.
16. Alcohol or drug abuse within the last 6 months
17. Use of medical marijuana
18. Use of recreational marijuana unless willing to undergo a 30-day washout prior to baseline
19. Use of any form of tobacco, including cigarette smoking, pipe smoking, or oral tobacco during the course of the trial; if a former smoker or tobacco user, the subject must not have used tobacco for 3 months before baseline
20. Consumes a low carbohydrate diet defined as less than 45% of total caloric intake as assessed by 7-day food record
21. Consumes MCT's, beta-hydroxybutyrate, other ketone supplements, coconut oil or palm kernel oil supplements, or goat milk products unless willing to undergo washouts
22. Current or recent use of oil supplements (fish oil, conjugated linoleic acid, etc.) unless willing to undergo specified washouts
23. Current or recent use of medications including drugs known to affect lipid or glucose metabolism unless willing to undergo washouts (e.g. steroids, beta-blockers, diuretics, insulin sensitizers, etc.)
24. Any other active or unstable medical condition, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant.
25. Blood donation 30 days prior to screening, during the study, or a planned donation within 30 days of the last study visit
26. Individuals who are cognitively impaired and/or who are unable to give informed consent
27. Participation in other clinical research trials one month prior to randomization will be assessed case-by-case by the QI

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Comparison of the change from baseline to day 30 between Brain Octane® Oil vs. placebo on reaction time as assessed by Dynavision D2 tests after first and second doses of Brain Octane® Oil | 30 days
  The Dynavision is a large, computerized light board with 64 buttons arranged in five concentric circles around an above-center, LCD display called the T-scope. The device allows for adjustable height and is adjusted for each participant such that the T-scope is approximately at eye level.The D2 version of the device connects to a laptop computer where results are displayed in a graph format, presenting individual progress. Participants will have their visual, motor, and physical reaction time measured using the Reaction Mode and Mode A on the Dynavision D2.
Comparison of the change from baseline to day 30 between Brain Octane® Oil vs. placebo on coordination as assessed by a Dynavision D2 test after first and second doses of Brain Octane® Oil | 30 days
  The Dynavision is a large, computerized light board with 64 buttons arranged in five concentric circles around an above-center, LCD display called the T-scope. The device allows for adjustable height and is adjusted for each participant such that the T-scope is approximately at eye level.The D2 version of the device connects to a laptop computer where results are displayed in a graph format, presenting individual progress. participants will have their coordination measured using the Mode A on the Dynavision D2.
Comparison of the change from baseline to day 30 between Brain Octane® Oil vs. placebo on the ability to perform cognitive tasks as assessed by a Dynavision D2 test and mod. Serial Sevens Test after first and second doses of Brain Octane® Oil | 30 days
  The Dynavision is a large, computerized light board with 64 buttons arranged in five concentric circles around an above-center, LCD display called the T-scope. The device allows for adjustable height and is adjusted for each participant such that the T-scope is approximately at eye level.The D2 version of the device connects to a laptop computer where results are displayed in a graph format, presenting individual progress. Participants will have their cognition measured using the Mode B on the Dynavision D2 device.
  The Serial Sevens Test was first introduced in the 1940's by Hayman for neurological examinations with regards to mental function in individuals with brain lesions. Over time, it has been modified and used to analyze cognitive function in healthy individuals.

SECONDARY OUTCOMES:
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in VO2Max (maximal oxygen consumption using cycle ergometer testing) as measured by Cardiocoach | 30 days
  The ergometer used will be an electromagnetically-controlled, stationary bicycle. Participants will use the ergometer in a temperature-controlled room, while intensity is incrementally increased. It will begin at 78W and increase by 39W every 3 minutes until volitional exhaustion by the participant. Participants will be instructed to maintain a cadence of 80 revolutions/min.
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in gas exchange threshold (GET, a measure of aerobic efficiency) as measured by Cardiocoach | 30 days
  The ergometer used will be an electromagnetically-controlled, stationary bicycle. Participants will use the ergometer in a temperature-controlled room, while intensity is incrementally increased. It will begin at 78W and increase by 39W every 3 minutes until volitional exhaustion by the participant. Participants will be instructed to maintain a cadence of 80 revolutions/min.
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in recovery from physical stress using Physical Fatigue Questionnaire | 30 days
  The Physical Fatigue Questionnaire uses a four-point scale to categorize physical fatigue. The scale ranges from zero (0) indicating no worse than usual to three (3) indicating much worse than usual. Individual question scores will be summed together to give a total score. A higher total score indicates more fatigue.
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in recovery from physical stress using Delayed Onset Muscle Soreness (DOMS) Questionnaire | 30 days
  The DOMS Questionnaire uses a seven-point scale to categorize muscle soreness. The scale ranges from one (1) indicating no pain to seven (7) indicating severe pain limiting the ability to move. Individual question scores will be summed together to give a total score. A higher total score indicates more DOMS.
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in acetoacetate plasma ketone measured before the first and second Dynavision tests | 30 days
  This will be analysed from blood samples.
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in beta-hydroxybutyrate plasma ketone measured before the first and second Dynavision tests | 30 days
  This will be analysed from blood samples.
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in glucose measured before first and second Dynavision D2 tests | 30 days
  This will be analysed from blood samples.
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in insulin measured before first and second Dynavision D2 tests | 30 days
  This will be analysed from blood samples.
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in creatine kinase measured before and after cycle ergometer testing | 30 days
  This will be analysed from blood samples.
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in fat body weight | 30 days
  Assess using bioelectrical impedance analysis (BIA)
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in percent body fat | 30 days
  Assess using bioelectrical impedance analysis (BIA)
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in lean dry mass | 30 days
  Assess using bioelectrical impedance analysis (BIA)
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in percent lean dry mass | 30 days
  Assess using bioelectrical impedance analysis (BIA)
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in total body water | 30 days
  Assess using bioelectrical impedance analysis (BIA)
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in percent body weight body water | 30 days
  Assess using bioelectrical impedance analysis (BIA)
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in basal metabolic rate | 30 days
  Assess using bioelectrical impedance analysis (BIA)

OTHER OUTCOMES:
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in the incidence of adverse events | 30 days
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in systolic blood pressure | 30 days
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in diastolic blood pressure | 30 days
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in heart rate | 30 days
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in complete blood count (CBC) in blood | 30 days
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in sodium levels in blood | 30 days
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in potassium levels in blood | 30 days
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in chloride levels in blood | 30 days
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in fasting glucose levels in blood | 30 days
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in creatinine levels in blood | 30 days
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in Aspartate Aminotransferase (AST) levels in blood | 30 days
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in Alanine Aminotransferase (ALT) levels in blood | 30 days
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in total bilirubin levels in blood | 30 days
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in total cholesterol levels in blood | 30 days
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in total low-density lipoprotein (LDL) levels in blood | 30 days
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in total high-density lipoprotein (HLDL) levels in blood | 30 days
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in triglyceride levels in blood | 30 days
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in NMR Lipoprotein levels in blood | 30 days
Comparison of the change from baseline to day 30 between Brain Octane® Oil versus placebo in Lp(a) levels in blood | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada